

## TRIAL STATISTICAL ANALYSIS PLAN

Document No.: c44527800-01

BI Trial No.: 1305-0039

Title: The effect of food on the pharmacokinetics of BI 1015550

(Formulation C2) following single oral dose administration in healthy subjects (an open-label, randomised, single-dose, two-

period, two-sequence crossover design)

(Revised Protocol including amendments 1&2 [c43335244-03]).

Investigational Product:

BI 1015550 (Nerandomilast)

Responsible trial statistician:

Phone:

Date of statistical 06 AUG 2024

Fax:

analysis plan:

Version: 1.0


Proprietary confidential information

© 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 1. TABLE OF CONTENTS

| TITLE P | 'AGE | 1 |
|---|---|---|
| 1. | TABLE OF CONTENTS | 2 |
| LIST OF | TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5.<br>5.1<br>5.2<br>5.2.1<br>5.2.2 | ENDPOINTS | 9<br>9<br>9 |
| 6.<br>6.1<br>6.2<br>6.3<br>6.4 | GENERAL ANALYSIS DEFINITIONS | 1<br>3<br>4 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS1 | 5 |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS1 | |
| 7. | PLANNED ANALYSIS | |
| 7.1<br>7.2 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS1 CONCOMITANT DISEASES AND MEDICATION1 | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY OBJECTIVE ANALYSIS2 | |
| 7.4.1 | Main analysis2 | |
| 7.5 | SECONDARY OBJECTIVE ANALYSIS2 | 2 |
| 7.5.1 | Key secondary objective analysis2 | |
| 7.5.2 | Secondary objective analysis2 | 2 |
| 7.5.2<br>7.7<br>7.8 | EXTENT OF EXPOSURE 2 SAFETY ANALYSIS 2 | 3 |
| 7.7 | EXTENT OF EXPOSURE | 3 |
| 7.7<br>7.8 | EXTENT OF EXPOSURE | 3<br>3<br>3 |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0039

Date: 06 AUG 2024, Version 1.0


05-0039 c44527800-01
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION28 |
|-----|-------------------------------------------------|
| 9. | REFERENCES29 |
| 10. | HISTORY TABLE30 |

# Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1305-0039


c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# LIST OF TABLES

| Table 6.1 | Treatments and labels used in the analysis | .11 |
|-------------|--------------------------------------------|-----|
| Table 6.4 | Subject sets analysed | .14 |
| Table 10: 1 | History table | .30 |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| ALT | Alanine Aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate Aminotransferase |
| $AUC_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| $\mathrm{AUC}_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BMI | Body mass index |
| BP | Blood pressure |
| CI | Confidence interval |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical trial plan |
| CTR | Clinical trial report |
| CV | Arithmetic Coefficient of Variation |
| DILI | Drug induced liver injury |
| EDMS | Electronic documentation management system |
| gCV | Geometric Coefficient of Variation |
| gMean | Geometric Mean |
| iPD | Important protocol deviations |
| Max | Maximum |
| Min | Minimum |
| N | Number non-missing observations |
| P10 | 10 <sup>th</sup> percentile |
| P90 | 90 <sup>th</sup> percentile |
| PKS | PK parameter analysis set |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| RPM | Report Planning Meeting |
| RAGe | Report Appendix Generator system |
| SD | Standard Deviation |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| Term | Definition / description |
|------|-----------------------------------|
| SOP | Standard Operating Procedure |
| TMF | Trial master file |
| TS | Treated Set |
| TSAP | P Trial Statistical Analysis Plan |
| ULN | Upper Limit of Normal |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 3. INTRODUCTION


As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

Study data (including data entered in the RAVE EDC system and external data provided by suppliers) will be stored in a Clinical Data Repository (CDR).

| Pharmacokinetic (PK) parameters will be calculated (version 8.1.1 or higher, version). | ulated using Phoenix WinNonlin <sup>TM</sup> software ) or SAS Version 9.4 (or later |
|---|---|
| The statistical analyses will be performed with including SAS <sup>TM</sup> (current Version 9.4, by of SAS <sup>TM</sup> -based tools (e.g., macros for the analyses) | ), and a number |
| Appendix Generator system (RAGe) for comp | ilation/formatting of the CTR appendices). |

c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

#### **Section 2.1.2 of the CTP:**

The following pharmacokinetic parameters will be determined for R-BI 1015550:

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

#### 5.2 SECONDARY ENDPOINTS

## 5.2.1 Key secondary endpoint

This section is not applicable as no key secondary endpoints have been defined in the CTP.

## 5.2.2 Secondary endpoint

#### Section 2.1.3 of the CTP:

The following pharmacokinetic parameter will be determined for R-BI 1015550:

•  $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)



## **Safety and tolerability endpoints**

#### Section 2.2.2.2 of the CTP:

Safety and tolerability of BI 1015550 will be assessed based on:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (blood pressure, pulse rate)
- Body weight

c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on treatments to be administered and selection of doses, refer to CTP Sections 3 and 4.

#### **Section 3.1 of the CTP:**


The trial will be performed as an open-label, randomised, single dose, two period, two-way crossover trial in healthy male and female subjects in order to compare the test treatment (T) to the reference treatment (R). [...] Subjects will be randomly allocated to the 2 treatment sequences (T--R or R-T). [...]

There will be a washout period of at least 10 days between the administrations of each treatment.

It is planned to include 18 healthy male and female subjects (at least 6 of each sex) in the trial.

For details of dosage and formulation see Table 6.1 below.

Table 6.1 Treatments and labels used in the analysis

| Treatment Treatment Short label group | | |
|---|---|---|
| R | BI 1015550, film-coated tablet, 18 mg, once, in fasting state | BI 18 mg fasted |
| T | BI 1015550, film-coated tablet, 18 mg, once, in fed state | BI 18 mg fed |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## Section 1.2.3 of the CTP:

. This is the period after the last dose during which measurable drug levels and/or pharmacodynamic effects are still likely to be present.

Based on this, the following study phases will be defined for the analysis of adverse events (AEs):

- Screening
  - Ranging from 0:00 h on day of informed consent until time of first drug administration.
- On treatment

- Ranging from the time of respective drug administration until (168 h) thereafter OR until next drug administration OR until trial termination (0:00 h on the day after trial termination), whatever occurs first.
- Follow-up (labelled "F/U")
  - Ranging from the end of REP until the next administration OR until trial termination (0:00 h on the day after trial termination), whatever occurs first.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### Section 7.2.5 of the CTP:

Note that AEs occurring after the last per protocol contact but entered before database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

The following AE displays will be provided in the Clinical Trial Report (CTR):

In Section 9.3 and Appendix 10.5.1.8 (for ClinicalTrials.gov and EudraCT) of the CTR displays, the on treatment phase will be analysed (labelled with the short label of the study treatment as in <u>Table 6.1</u>). The screening and follow-up phases will not be included in this analysis.

The following totals will be provided in addition for AE outputs for Section 9.3:

• A total over all on treatment phases ("Total")

In Section 9.4 and Appendix 10.6 (Listings) of the CTR displays, the screening period, as well as the follow-up phases will additionally be included. The labelling of the actual treatment in listings corresponds to the labelling of study phases defined above. Single exception is the Follow-up phase where the actual treatment will be labelled "F/U <short label>".

For detailed information on the handling of the treatments refer to Technical TSAP ADS (analysis data set) plan and Analysis Data Reviewers guide.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all treated subjects. Consistency check listings (for identification of deviations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting (RPM). At this meeting, all manual deviations identified at the sites by the CRAs and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPD), and for the process of identification of these, refer to the Boehringer Ingelheim (BI) SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

Important protocol deviation (iPD) categories are pre-specified in the iPD specification file (DV domain) (3). IPDs will be identified no later than in the RPM, and the iPD categories will be updated as needed.

If any iPDs are identified, they are to be summarised into categories and will be captured in the iPD specification file (DV domain) (3) and in the decision log (4). Both documents will be stored within the TMF in EDMS.

The iPDs will be summarized and listed in the CTR.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## **6.3 INTERCURRENT EVENTS**

This section is not applicable.

## 6.4 SUBJECT SETS ANALYSED

#### Section 7.2.1.1 of the CTP:

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were treated with at least one dose of trial drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model-based analyses of PK parameters will be based on the PKS.

Table 6.4 Subject sets analysed

| | Subject analysis set | |
|-----------------------------------------|----------------------|-----|
| Class of analysis/endpoint | TS | PKS |
| Primary and secondary endpoints | | X |
| | | X |
| Safety assessments | X | |
| Disposition | X | |
| Demographics / baseline characteristics | X | |
| Important protocol deviations | X | |
| Exposure | X | |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.3:

It is not planned to impute missing values for safety parameters.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see "Handling of Missing and Incomplete AE Dates") (5).

Missing data and outliers of PK data are handled according to BI standards (see "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics" (6) and "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (7)).

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

## Section 7.2.5 of the CTP:

For laboratory data and vital signs, baseline is defined as measurement prior to first drug administration.

#### **Section 6.1 of the CTP:**


Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and the end of study examination are provided in the CTP Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration.

If not stated otherwise in the CTP Flow Chart, the acceptable deviation from the scheduled time for vital signs, ECG, and laboratory tests will be  $\pm$  30 min.

If scheduled in the CTP Flow Chart at the same time as a meal, blood sampling, vital signs, and 12-lead ECG recordings have to be done first. Furthermore, if several measurements including venipuncture are scheduled for the same time, venipuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the CTP Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

The acceptable deviations from the nominal blood sampling times are as follows:

• The pre-dose samples will be taken  $\leq 3h$  before dosing.

c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

- 0 to 2 h post-dose samples will be taken within  $\pm$  2 min of the planned post-dose sampling time.
- 2.5 to 4 h post-dose samples will be taken within  $\pm$  5 min of the planned post-dose sampling time.
- 6 to 12 h post-dose samples will be taken within  $\pm$  10 min of the planned post-dose sampling time.
- 24 h or later post-dose samples will be taken within  $\pm$  60 min of the planned post-dose sampling time.

If a subject misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

Unscheduled measurements of laboratory data and vital signs data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 7. PLANNED ANALYSIS

Safety analysis (refer to Section 7.8) will be performed by will be presented in Sections 9.1 to 9.4 of the CTR and in Appendix 10.6 and 10.5.1.

Inferential statistical analyses of PK endpoints (refer to Section 7.4) will also be performed by and will be presented in Section 9.5 of the CTR and in Appendix 10.5.3.

Descriptive data analysis of PK endpoints and concentrations will be performed by the and will be presented in Section 9.6 of the CTR and in Appendix 10.5.5.

The format of the listings and tables will follow the BI standards (see "Standards for Reporting of Clinical Trials and Project Summaries" (8)) with the exception of those generated for PK-calculations following BI standards for PK/PD analysis (9).

The individual values of all subjects will be listed, sorted by treatment sequence, subject number, visit and time point. The listings will be included in Appendix 10.6 of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations and PK parameters, the following descriptive statistics will additionally be calculated (if needed):

Nobs number of observations

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile


The data format for descriptive statistics of concentrations will be identical to the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The gMeans and gMean ratio based on the inferential statistics will be reported with maximum of 2 decimal places.

Tabulations of frequencies for categorical data will include all possible categories available in the CRF and will display the number of observations in a category, as well as the percentage (%). Percentages will be given in integer numbers due to the small sample size of <100. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in brackets (e.g. (mg)).

## Exclusion of PK parameters

The ADS "ADPP" (PK parameters) contains column variables APEX and APEXCO indicating inclusion/exclusion (APEX) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters only if they are not flagged for exclusion, that is APEX is equal to "Included".

## Exclusion of PK concentrations


The ADS "ADPC" (PK concentrations per time-point or per time-interval) contains column variables ACEX and ACEXCO indicating inclusion/exclusion (ACEX) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to

- 'ALL CALC', the value will be excluded for all types of analyses based on concentrations.
- 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval.
- 'HALF LIFE', the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda_z$ ) only; the value is included for all other analyses.

If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (7) and "Description of Analytical Transfer Files and PK/PD Data Files" (10).

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR, based on the TS. The data will be summarised by the treatment sequence and in total.

## 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the CTR, based on the TS.

Concomitant diseases and non-drug therapies will be coded according to the version defined in the decision log (4) of the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Concomitant medications will be coded according to the most recent version of the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

In the remaining document 'therapy' will be used for non-drug therapies and concomitant medications.

#### Section 7.2.5 of the CTP:


Previous and concomitant therapies will be presented per treatment without consideration of actual period.

The diagnoses and therapies will be listed. Subjects without any concomitant diagnoses or concomitant therapies will be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK data will be decided no later than at the RPM.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 7.3 TREATMENT COMPLIANCE


Treatment compliance will not be analysed as a specific endpoint, but judged by observed analyte concentrations, cf. **Section 4.3 of the CTP:** 

Compliance will be assured by administration of all trial medication in the trial centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

Any deviations from complete drug intake will be addressed in the RPM and described in the CTR.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.4 PRIMARY OBJECTIVE ANALYSIS

Independent of the main objectives stated in the CTP, this section describes further details of the primary endpoint analyses outlined in the CTP.

### 7.4.1 Main analysis

#### Section 7.2.2 of the CTP:

The primary endpoints (refer to CTP Section 2.1.2) will be calculated with Non-Compartmental Analysis (NCA).

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{ijkm} = \mu + \zeta_i + s_{im} + \pi_j + \tau_k + e_{ijkm}$$
 where

 $y_{ijkm}$ = logarithm of response measured on subject m in sequence i receiving treatment k in period j,

μ the overall mean,

 $\zeta_i$  the  $i^{th}$  sequence effect, i = 1, 2

 $s_{im}$  the effect associated with the  $m^{th}$  subject in the  $i^{th}$  sequence,  $m=1, 2, ..., n_i$ 

 $\pi_j$  the  $j^{th}$  period effect, j = 1, 2

tk the  $k^{th}$  treatment effect, k = 1, 2

 $e_{ijkm}$  the random error associated with the  $m^{th}$  subject in sequence i who received treatment k in period j.

where  $s_{im} \sim N(0, \sigma_B^2)$  i.i.d.,  $e_{ijkm} \sim N(0, \sigma_W^2)$  i.i.d. and  $s_{im}$ ,  $e_{ijkm}$  are independent random variables.

Point estimates for the ratios of the geometric means (Test/Reference) for the primary endpoints (see CTP Section 2.1) and their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

The implementation for this analysis will be accomplished by using the CSD macros based on the PKS. The following SAS code can be used:

PROC MIXED DATA=indata METHOD=REML;


CLASS subject treatment sequence period;

MODEL logpk = treatment sequence period / DDFM=KR;

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

RANDOM subject(sequence); LSMEANS treatment / PDIFF CL ALPHA=0.1;

RUN;



## 7.5 SECONDARY OBJECTIVE ANALYSIS

Independent of the main objectives stated in the CTP, this section describes further details of the secondary endpoint analyses.

## 7.5.1 Key secondary objective analysis

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 Secondary objective analysis

## Section 7.2.3 of the CTP:


The secondary endpoints (refer to CTP Section 2.1.3) will be calculated with NCA and will be assessed statistically using the same methods as described for the primary endpoints.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



#### Safety endpoints

For a description of the analysis of safety and tolerability, please refer to Section 7.8.

#### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available.

**Section 7.2.5 of the CTP:** For all analyses, the treatment actually administered (= treatment at onset) to the subject will be used (any deviations from the randomised treatment will be discussed in the minutes of the Report Planning Meeting).

## 7.8.1 Adverse Events


AEs will be coded using MedDRA. The coding version number will be displayed as a footnote in the respective output.

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs. BI standards as presented in "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template" [BI-KMED-BDS-HTG-0041] (11) and [BI-KMED-BDS-HTG-0066] (12) will be applied.


c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to 'screening', 'on-treatment' or 'follow-up' phases as defined in Section 6.1. AEs will be analysed based on actual treatments, as defined in Table 6.1.

An overall summary of adverse events will be presented. This overall summary will comprise summary statistics for the class of AESIs.

### Section 5.2.6.1.4 of the CTP:

The following are considered as AESIs:

### • Potential severe DILI

A potential severe Drug Induced Liver Injury (DILI) that requires follow-up is defined by the following alterations of hepatic laboratory parameters:

- 1. AST (aspartate aminotransferase) and/or ALT (alanine aminotransferase) elevation  $\geq 3x$  ULN and TB (total bilirubin)  $\geq 2x$  ULN measured at the same visit, or in samples drawn within 30 days of each other, OR
- 2. AST and/or ALT elevation  $\geq 3x$  ULN and INR  $\geq 1.5x$  ULN measured at the same visit, or in samples drawn within 30 days of each other, OR
- 3. AST and/or ALT elevation  $\geq 3x$  ULN with new onset, or worsening of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%), OR
- 4. AST and/or ALT elevation  $\geq 5x$  ULN [...]

### • Vasculitis events


In this CTP, vasculitis is defined as any event term included in the MedDRA SMQ Vasculitis (broad). This includes clinical and pathological features related to primary or secondary vasculitis syndromes and involving any type, size, and location of blood vessels. [...]

• Serious infections, opportunistic or mycobacterium tuberculosis infections [...]

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (13), in addition to Deaths and serious adverse events, 'other significant' AEs need to be listed in the CTR. These will be any non-serious adverse event that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted).

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with serious AEs, for subjects with investigator-defined drug-related AEs, for subjects with investigator-defined drug-related serious adverse events, for subjects with AESIs and for subjects with AEs leading to discontinuation. In addition, the frequency of subjects with AEs will be summarised by worst intensity, treatment, primary system organ class (SOC) and preferred term (PT).

c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The system organ classes will be sorted by default alphabetically, PTs will be sorted by descending frequency (within SOC).

In addition, for disclosure of AE data on ClinicalTrials.gov, frequencies of subjects with non-serious AEs that had an incidence of > 5% (in preferred terms) for at least one treatment will be summarised by treatment, primary SOC and PT. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs and the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards [BI-KMED-BDS-HTG-0042] (14). Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

**Section 7.2.5 of the CTP**: Laboratory data will be compared to their reference ranges. Values outside the reference range will be highlighted in the listings. Additionally, differences from baseline will be evaluated.

It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Clinically significant abnormal laboratory values are identified either in the Investigator's comments or at the Report Planning Meeting at the latest. They will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment).

For post-dose measurements of laboratory data, descriptive statistics including change from baseline will be calculated by planned time point based on the first value of the subject at that planned time point (or assigned to that planned time point). For baseline value, the measurement before first drug administration will be used.

### 7.8.3 Vital signs


Descriptive statistics over time including change from baseline will be performed for vital signs (blood pressure and pulse rate) and body weight. In the listing the change from baseline will also be displayed. In addition, the time profiles of median (Min, Max) will be displayed graphically by treatment group.

For post-dose measurements of vital signs, descriptive statistics will be calculated by planned time point based on the first value of the subject at that planned time point (or assigned to that planned time point). For baseline value, the measurement before first drug administration will be used.

Clinically relevant findings in vital signs will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such.

c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



c44527800-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be loaded into the trial database during trial conduct in accordance with the open label fashion of the trial as described in the CTP section 4.1.5.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 9. REFERENCES

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | BI-VQD-12045_40-413: "Identify and Manage Important Protocol Deviations (iPD)", current version, Group "Clinical Operations", KMED. |
| 3. | <i>BI-KMED-BDS-TMP-0059</i> : "iPD specification document (sdtm-dv-domain-specification)", template, current version, Group "Clinical Operations", KMED. |
| 4. | 001-MCS-50-415_RD-03: "Clinical Trial Analysis Decision Log (template)", current version, Group "Biostatistics & Data Sciences", KMED. |
| 5. | <i>BI-KMED-BDS-HTG-0035:</i> "Handling of Missing and Incomplete AE Dates", current version, Group "Biostatistics & Data Sciences" KMED. |
| 6. | <i>BI-KMED-TMCP-HTG-0025:</i> "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version;, Group "Translational Medicine Clinical Pharmacology", KMED. |
| 7. | <i>BI-KMED-TMCP-MAN-0014:</i> "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| 8. | BI-KMED-BDS-HTG-0045: "Standards for Reporting of Clinical Trials and Project Summaries", current version, Group "Biostatistics & Data Sciences", KMED. |
| 9. | <i>BI-KMED-TMCP-OTH-0003</i> : "Graphs and Tables for Clinical Pharmacokinetics and Pharmacodynamic Noncompartmental Analyses", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| 10. | <i>BI-KMED-TMCP-MAN-0010</i> : "Description of Analytical Transfer Files and PK/PD Data Files", current version, Group "Translational Medicine Clinical Pharmacology", KMED. |
| 11. | <i>BI-KMED-BDS-HTG-0041</i> : "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template", current version, Group "Biostatistics & Data Sciences", KMED. |
| 12. | BI-KMED-BDS-HTG-0066: "Analysis and Presentation of AE data from clinical trials", current version, Group "Biostatistics & Data Sciences", KMED. |
| 13. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version, EMA webpage. |
| 14. | BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version, Group "Biostatistics & Data Sciences", KMED. |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 10. HISTORY TABLE

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1.0 | 06-AUG-24 | | None | This is the final TSAP. |